CLINICAL TRIAL: NCT06735365
Title: Comparative Effectiveness of Oxiris Filters Versus Conventional Hemofilters in Septic Patients: a Retrospective Cohort Study
Brief Title: Comparative Effectiveness of Oxiris Hemofilters Versus Conventional Hemofilters in Septic Patients
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-05-02
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Sepsis - to Reduce Mortality in the Intensive Care Unit; Hemodiafiltration; Cytokine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Oxiris: The group which we used oxiris filter for CRRT.
  Interventions: Other: CRRT
- Non-Oxiris: The group which we used other filters like M150 for CRRT.
  Interventions: Other: CRRT

INTERVENTIONS:
Other: CRRT — Hemodiafiltration

SUMMARY:
We divided patients in 2 groups. First group was the patients who received Oxiris filters during CRRT. Second group was the patiens who have received CRRT filters other than Oxiris.

We compared the lab parameters (Urea, Creatinin, Lactate, ABG parameters and SOFA escore with together.

ELIGIBILITY:
Inclusion Criteria:

sepsis diagnosis CRRT indication

Exclusion Criteria:

patients under age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study population includes patients who have admission on our clinic for more than 5 days and diagnosed with sepsis who has CRRT indication
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
SOFA Score | 6 month
  We compared SOFA scores of patients on admission and on 5th day.

SECONDARY OUTCOMES:
Survival comparison | 6 month
  We compared patients survival rates between two group.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr Sadi Konuk Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No